CLINICAL TRIAL: NCT00207831
Title: Trial UFT/RT Randomized Multicenter Phase III Randomized Trial Testing Ftorafur (UFT) Associated With Neoadjuvant Radiotherapy Versus Radiotherapy Alone in Rectal Adenocarcinoma
Brief Title: Trial Testing Ftorafur (UFT) Associated With Neoadjuvant Radiotherapy Versus Radiotherapy Alone in Rectal Adenocarcinoma
Acronym: UFT RT Phase 3
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Terminated after interim analysis
Sponsor: Institut Cancerologie de l'Ouest (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CPP276
Record Dates: First submitted 2005-09-13; First posted 2005-09-21 (Estimated); Last update posted 2020-03-25 (Actual); Status verified 2020-03

CONDITIONS: Rectal Cancer; Stage II/III; T3 or T4 (Only Anal Extension) Rectal Cancer; N0-2; M0
Keywords: rectal cancer; neoadjuvant therapy; UFT; radiochemotherapy
MeSH Terms: conditions — Rectal Neoplasms | interventions — Tegafur; Uracil

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Tegafur uracile + radiotherapy (Experimental)
  Interventions: Drug: Tegafur and Uracil
- radiotherapy (Active Comparator)
  Interventions: Drug: Tegafur and Uracil

INTERVENTIONS:
Drug: Tegafur and Uracil

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as 5-fluorouracil, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing and also as a radiosensibilisant. Radiation therapy uses high-energy x-rays to kill tumor cells. 5-fluorouracil may make tumor cells more sensitive to radiation therapy. Oral 5-fluorouracil is more convenient for ambulatory patients. Giving UFT (Tegafur and Uracil) with radiation therapy before surgery may shrink the tumor so it can be removed.

PURPOSE: This phase III trial is studying how well giving UFT with radiation therapy works in treating patients who are undergoing surgery for operable rectal cancer.

DETAILED DESCRIPTION:
Adenocarcinoma of the rectum

Stage II/stage III rectal cancer (if T4 only anal extension eligible)

Drug: UFT

Procedure: chemotherapy

Procedure: conventional surgery

Procedure: neoadjuvant therapy

Procedure: radiation therapy

Procedure: radiosensitization

Procedure: surgery

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed invasive adenocarcinoma of the rectum , M0, lower side < 10 cm from anal verge
* T3 or T4 disease (T4 exclusive anal extension )

PATIENT CHARACTERISTICS:

Performance status

* ECOG 0-2 OR
* Zubrod 0-2

Life expectancy

* Not specified

Hematopoietic

* Absolute neutrophil count > 1,500/mm^3
* Platelet count ≥ 100,000/mm^3

Hepatic

* Bilirubin < x2 UNL

Renal

* Creatinine < 150 µMol/L

Gastrointestinal

* No history of inflammatory bowel disease
* No history of difficulty or inability to take or absorb oral medications

Neurologic

* Not specified

Other

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No other malignancy within the past 5 years except curatively treated basal cell skin cancer or carcinoma in situ of the cervix
* No history of psychiatric conditions or diminished mental capacity that would preclude study compliance or giving informed consent

PRIOR CONCURRENT THERAPY:

Chemotherapy

* No prior chemotherapy

Radiotherapy

* No prior radiotherapy to the pelvis

Other

* No other concurrent investigational drugs
* No other concurrent anticancer treatment

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 219 (Actual)
Dates: Start 2004-07 (Actual); Primary Completion 2007-06 (Actual); Study Completion 2008-02 (Actual)

PRIMARY OUTCOMES:
Compare the rate of pathologic complete response of the primary tumor in patients with operable rectal cancer receiving preoperative chemoradiotherapy versus patients receiving radiotherapy alone

SECONDARY OUTCOMES:
Compare endoscopic ultrasonographic response in patients with operable rectal cancer receiving preoperative chemoradiotherapy versus patients receiving radiotherapy alone.
Compare quality of life (Quality of Life Questionnaire Core 30 Items [QLQ-C 30])
Compare the rate of sphincter conservation alone.
Compare the safety of the chemoradiotherapy regimen to radiotherapy alone
Compare the rate of resectability with negative resection margins in patients treated with this two regimen.
Compare recurrence free survival and disease free survival
Compare overall survival

CONTACTS AND LOCATIONS:
Overall Officials: Patrice Cellier, MD, Study Chair — Institut Cancerologie de l'Ouest; Rémy Barraya, MD, Study Chair — Institut Cancerologie de l'Ouest; Christian Chevelle, MD, Study Chair — Centre des Hautes Energie, Toulouse; Gérard Lorimier, MD, Study Chair — Institut Cancerologie de l'Ouest; Véronique Verrièle, MD, Study Chair — Institut Cancerologie de l'Ouest; Michèle Boisdron, Pct, PhD, Study Chair — Institut Cancerologie de l'Ouest; Loïc Campion, MD, Study Chair — Centre René Gauducheau, Nantes
Locations (27):
- France (27):
  - Clinique Sainte Catherine, Avignon
  - Hopital Avicenne, Bobigny
  - Institut de Cancérologie et d'Hématologie, Brest
  - Centre Hospitalier, Brive-la-Gaillarde
  - Centre d'Oncologie-radiothérapie d'Eure et Loir, Chartres
  - Centre Jean Perrin, Clermont-Ferrand
  - Centre Médical République, Clermont-Ferrand
  - Clinique du Mail, Grenoble
  - Centre Hospitalier Départemental, La Roche-sur-Yon
  - Centre Guillaume le Conquérant, Le Havre
  - Centre Oscar Lambret, Lille
  - Centre Hospitalier, Lorient
  - Centre léon Bérard, Lyon
  - Centre Gray, Maubeuge
  - Clinique du Pont de Chaume, Montauban
  - Polyclinique St Roch, Montpellier
  - Centre Hospitalier, Niort
  - Clinique Valdegour, Nîmes
  - Centre Hospitalier Universitaire, Poitiers
  - Centre Hospitalier de Cornouaille, Quimper
  - Centre Eugène Marquis, Rennes
  - Centre Hospitalier, Rodez
  - Centre Frédéric Joliot, Rouen
  - Clinique Armoricaine de Radiologie, Saint-Brieuc
  - Centre de Radiothérapie, Strasbourg
  - Centre des Hautes Energies, Toulouse
  - Clinique Fleming, Tours